CLINICAL TRIAL: NCT04297527
Title: Efficacy of Mulligan Mobilization Technique in Chronic Non-Spesific Low Back Pain
Brief Title: Effect of Mulligan Mobilization in Chronic Non-Spesific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Şule, Lecturer, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.11.2016/20
Record Dates: First submitted 2020-02-24; First posted 2020-03-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Chronic Pain
Keywords: Lumbal SNAGs, efficiency
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator
Masking Description: All assessments were made by another blind researcher three times at before, after and 6 month after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy Group (Experimental): Group I (18 subjects) received 15 sessions of Conventional Physiotherapy program (CPP) 5 times per week.
  Interventions: Procedure: Conventional Physiotherapy
- Mulligan Mobilization Group (Experimental): Mulligan Mobilization was administered 9 sessions (3 days a week, for 3 weeks). .
  Interventions: Procedure: Mulligan Mobilization
- Conventional Physiotherapy plus Mulligan Mobilization Group (Experimental): Conventional Physiotherapy (15 session) plus Mulligan Mobilization Programme (9 session) were applied in this group. CP were applied 5 days a week and CP+MM 3 days a week for 3 weeks.
  Interventions: Procedure: Conventional Physiotherapy; Procedure: Mulligan Mobilization

INTERVENTIONS:
Procedure: Conventional Physiotherapy — Conventional Physiotherapy consist of Hotpacks, TENS and US.The participants were positioned in prone and supported with a pillow under the abdomen, 20 min hot pack was applied. Therapatic Ultrason were applied with the frequency of 1 MHz, intensity of 1,5 watt/cm² and duration of 5 minute. TENS was applied to the lumbar region with 2-channel, 4 surface electrodes at 60-120 Hz, and 50-100 pulse duration for 20 minutes.
  Arms: Conventional Physiotherapy Group; Conventional Physiotherapy plus Mulligan Mobilization Group
Procedure: Mulligan Mobilization — Extension SNAGS in prone, SNAGS in lion position and Lumbar flexion SNAGS in sitting, techniques were used. The techniques were applied in 3 sets with 10 repetitions and 60 seconds rest between sets.
  Other Names: Lumbal SNAGs
  Arms: Conventional Physiotherapy plus Mulligan Mobilization Group; Mulligan Mobilization Group

SUMMARY:
Fifty five participants diagnosed with CNSLBP, will randomized into three groups. Group I (18 subjects) will receive 15 sessions of Conventional Physiotherapy program (CPP) 5 times per week, Group II (19 subjects) will receive 9 sessions of SNAGs, and Group III will receive CPP plus SNAGs. Outcome measures are pain, ROM, spinal mobility, fear avoidance behaviour and function. Measurements will record before, after and 6 month after the end of the treatment.

DETAILED DESCRIPTION:
Inclussion criterias are; low back pain for at least 3 months, intensity of pain ranges from 3 to 6 according to VAS. Exclussion criterias are; undergoing surgical operation in the lumbar region or having a surgical indication, having an exercise therapy and / or physical therapy in the last 1 year, a history of trauma involving lumbar region and systemic and inflammatory disease targeting this region, participants using corticosteroids for a long time and being pregnant.Acording to our criterias 55 participants diagnosed with CNSLBP will randomised into three groups. Group 1 will receive Conventional Physiotherapy programme consisting of Hot pack, US and TENS applications. Group II aill receive Lumbar SNAGS consisting of Lumbar Extension SNAGS in prone, SNAGS in lion position and Lumbar flexion SNAGS in sitting, techniques. Group III will receive 9 sessions of SNAGs, and Group III will receive CPP plus SNAGs.Outcome measures are pain, ROM, spinal mobility, fear avoidance behaviour and function. Measurements will record before, after and 6 month after the end of the treatment. All treatment groups were treated with the same researcher. All assessments were made by another blind researcher three times at before, after and 6 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* low back pain for at least 3 months
* intensity of pain ranges from 3 to 6 according to VAS

Exclusion Criteria:

* undergoing surgical operation in the lumbar region or having a surgical indication having an exercise therapy and / or physical therapy in the last 1 year
* a history of trauma involving lumbar region and systemic and inflammatory disease targeting this region
* corticosteroids consumption for a long time
* being pregnant.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Change of Range of Motion from baseline at 3 weeks and from baseline at 6 months | Baseline, 3 weeks,6 months
  ROM is measured by BROM II device during flexion and extension activity.
Change of Spinal Mobility from baseline at 3 weeks and from baseline at 6 months | Baseline, 3 weeks,6 months
  Spinal mobility measured by Schober test.
Change from Pain Intensity from baseline at 3 weeks and from baseline at 6 months | Baseline, 3 weeks,6 months
  Pain intensity during flexion and extension activity in lumbar region is measured by Numeric pain scale in which "0" shows No pain while "10" shows worst pain.

SECONDARY OUTCOMES:
Change from Fear Avoidance Behaviour from baseline at 3 weeks and from baseline at 6 months | Baseline, 3 weeks,6 months
  It ıs measured by Fear Avoidance Behaviour Questionnaire-Turkish.The total score ranges from 0 to 96. Maximum score indicates increased fear avoidanve behaviour
Change from Disability level from baseline at 3 weeks and from baseline at 6 months | Baseline, 3 weeks,6 months
  It ıs measured by measured by Rolland Morris Disability Questionnaire-Turkish.Total score ranked from 0 to 24. İncreased score represents disability in functional activities

CONTACTS AND LOCATIONS:
Overall Officials: Nesrin Yağcı, Prof. Dr., Study Director — Pamukkale University
Locations (1):
- Denizli State Hospital, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because there is no web site to share my data

REFERENCES:
- [Background] Hidalgo B, Pitance L, Hall T, Detrembleur C, Nielens H. Short-term effects of Mulligan mobilization with movement on pain, disability, and kinematic spinal movements in patients with nonspecific low back pain: a randomized placebo-controlled trial. J Manipulative Physiol Ther. 2015 Jul-Aug;38(6):365-74. doi: 10.1016/j.jmpt.2015.06.013. Epub 2015 Jul 26. PMID 26215900
- [Background] Vicenzino B, Paungmali A, Teys P. Mulligan's mobilization-with-movement, positional faults and pain relief: current concepts from a critical review of literature. Man Ther. 2007 May;12(2):98-108. doi: 10.1016/j.math.2006.07.012. Epub 2006 Sep 7. PMID 16959529
- [Background] Hussien HM, Abdel-Raoof NA, Kattabei OM, Ahmed HH. Effect of Mulligan Concept Lumbar SNAG on Chronic Nonspecific Low Back Pain. J Chiropr Med. 2017 Jun;16(2):94-102. doi: 10.1016/j.jcm.2017.01.003. Epub 2017 Mar 30. PMID 28559749